CLINICAL TRIAL: NCT00449436
Title: A Randomised, Open-Label Study to Evaluate the Efficacy and Safety of a Treatment Optimisation With Trizivir During 96 Weeks After a First Antiretroviral Treatment in HIV-1 Infected Subjects.
Brief Title: Study To Evaluate Long Term Maintenance With TRIZIVIR After Boosted Protease Inhibitor (PI) Or Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI) In HIV-1 Infected Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 103441
Record Dates: First submitted 2007-03-19; First posted 2007-03-20 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: HIV Infections
Keywords: treatment experienced; HIV
MeSH Terms: conditions — HIV Infections | interventions — abacavir, lamivudine, and zidovudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: TRIZIVIR — TRIZIVIR
Drug: Non-nucleoside reverse transcriptase inhibitor — Non-nucleoside reverse transcriptase inhibitor
Drug: Boosted Protease Inhibitor — Boosted Protease Inhibitor
  Other Names: TRIZIVIR; Non-nucleoside reverse transcriptase inhibitor

SUMMARY:
The current goal of antiretroviral therapy is to use a potent regimen that will suppress plasma viral load and maintain this suppression as long as possible. However, for most patients treated with such potent regimen, several problems can limit their long term effectiveness and contribute to incomplete viral suppression. These problems include poor tolerability, metabolic toxic effects. In order to avoid common problems as toxicity it might be interested to simplify treatment with fewer toxicity, lower pill burden. In this study we will evaluate the safety and efficacy of a simplification treatment with TRIZIVIR in long term after a Boosted PI or NNRTI containing regimen as first line therapy.

ELIGIBILITY:
Inclusion criteria:

* Subject is ≥18 years of age and has documented evidence of HIV-1 infection.
* Patient received first-line therapy including a boosted Protease Inhibitor or NNRTI for at least 6 months. Note: Only the patients whose first line antiretroviral treatment was modified for intolerance (and not for virological failure) could be included provided this treatment has been stable for at least 6 months.
* Patient having a viral load < 50 copies/ml at screening and at least 3 months prior to enrollment,
* Subject is willing and able to understand and provide written informed consent prior to participation in this study.
* For women of childbearing potential: has a negative pregnancy test result (-human chorionic gonadotropin; -HCG) within 35 days prior to administration of investigational product (Day 1) and agrees to use a proven double barrier method of contraception or abstinence from 2 weeks before the first day of treatment.

Exclusion criteria:

* Patient has received Trizivir®.
* Patient has a viral load > 50 copies/mL at the screening and within 3 months of enrollment.
* Patient has one or more CDC (1993) category C events in acute phase in classification of infection HIV.
* Grade 3 ALT, AST (between 5 and 10 times normal higher limit) or Grade 4 (more than 10 times normal higher limit) for the during screening and before the first day of treatment (1-28 days);
* Presence clinically-relevant of pancreatitis or hepatitis within 6 months of screening;
* Patient has a severe hepatic insufficiency or a renal insufficiency in final stage.
* Any situation (such as for example drug-addiction or active alcoholism) which, of the opinion of the investigator, could interfere with the observance and the evaluations required by the protocol and which could compromise the safety of the patient during his participation in the study;
* Pregnancy, nursing, or pre-menopausal woman likely to be pregnant and not receiving reliable contraception (oral contraception, progesterone injectable associated a mechanical method of protection, intra-uterine device...) for the duration of study
* Any biological anomaly for the period of the study and before the first day of treatment which, of the opinion of the investigator, could contra-indicate the participation of the patient in the study. Any biological anomaly of Grade 4 for the period of study and before the first day of treatment , except contrary opinion of the investigator and after agreement of the sponsor;
* Any pathological state (diabetes, hyperthyroidism, syndrome of malabsorption, renal insufficiency...) which, of the opinion of the investigator, could interfere on absorption, the distribution, the metabolism and the excretion of the drugs;
* Onset of allergy to the drugs of the study or other allergies which, of the opinion of the investigator, contra-indicates the participation of the patient in the study;
* Patient is taking part in a clinical trial at the time of entry in the study except for observational trials.
* Treatment by an experimental drug in the 30 days or five half-lives of the treatment (the longest period will be taken) which precede the first treatment of the test. (After opinion of the sponsor.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2005-01-10 (Actual); Primary Completion 2007-12-12 (Actual); Study Completion 2007-12-13 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a HIV plasma RNA<50 copies/ml at 48 weeks | 48 weeks
  Proportion of patients with a HIV plasma RNA<50 copies/ml at 48 weeks

SECONDARY OUTCOMES:
Proportion of patients with a HIV plasma RNA <50copies/ml at 96 weeks. | up to 96 weeks
  Proportion of patients with a HIV plasma RNA <50copies/ml at 96 weeks
CD4 count profile at baseline 24 W,48 and 96 W | 24, 48, 96 weeks
  CD4 count profile at baseline 24,48, and 96 weeks
Genotypic profile resistance | up to 96 weeks
  Genotypic profile resistance
Determination of compliance of patient to treatment | up to 96 weeks
  Determination of compliance of patient to treatment
Proportion of patients having a viral load <50 copies/mlL at 96 weeks in the ITT (M=F) population; | up to 96 weeks
  Proportion of patients having a viral load <50 copies/mlL at 96 weeks in the ITT (M=F) population
Proportion of patients with a virl load <50 copies/mL at 96 weeks (per protocol population) | up to 96 weeks
  Proportion of patients with a viral load <50 copies/mL at 96 weeks (per protocol population)
Proportion of patients with a viral load <5 copies/mL at 96 weeks | up to 96 weeks
  Proportion of patients with a viral load <5 copies/mL at 96 weeks
Change from baseline in CD4 counts at 24, 48, 96 weeks; Genotypic resistance profile of the HIV-1 in the event of virological failure CV >1000 copies/mL, as confirmed twice; Time to virologic failure (by Kaplan - Meier) | 24, 48, 96 weeks
  Change from baseline in CD4 counts at 24, 48, 96 weeks; Genotypic resistance profile of the HIV-1 in the event of virological failure CV >1000 copies/mL, as confirmed twice; Time to virologic failure (by Kaplan - Meier)
Patient adherence (using the PMAQ3 instrument); Retrospective determination of HLAB57 as a marker for hypersensitivity reaction in patients randomized to the Trizivir arm. | up to 96 weeks
  Patient adherence (using the PMAQ3 instrument); Retrospective determination of HLAB57 as a marker for hypersensitivity reaction in patients randomized to the Trizivir arm.
Quantitative measurement of the residual replicative capacity (using cell-based assay) using number of quiescent cells and quantification of proviral DNA. | up to 96 weeks
  Quantitative measurement of the residual replicative capacity (using cell-based assay) using number of quiescent cells and quantification of proviral DNA.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline